CLINICAL TRIAL: NCT05606341
Title: Phase 1 Clinical Trial of Innate Immunity Stimulation Via TLR9 in Early Alzheimer's Disease (AD)
Brief Title: Innate Immunity Stimulation Via TLR9 in Early AD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20-00267
Record Dates: First submitted 2022-11-01; First posted 2022-11-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment; Alzheimer Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — 1018 oligonucleotide

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly allocated in a blinded fashion to receive s.c. injection of either CpG ODN (dose level 1, 0.1 mg/kg) or placebo (saline). Dose escalation will occur after 10 weeks after the last injection in a new subject cohort, and will be based on the safety data and immunostimulatory assessments at previous dose level cohorts.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CpG 1018 0.1 mg/kg (Experimental): 3 injections at Day 1, Week 4, and Week 8.
  Treatment administered as morning injection of dose 0.1mg/kg, followed by 1-hour post-dose observation period to check for injection site reaction and/or adverse reactions.
  Interventions: Drug: CpG1018
- CpG 1018 0.25 mg/kg (Experimental): 3 injections at Day 1, Week 4, and Week 8.
  Treatment administered as morning injection of dose 0.25 mg/kg, followed by 1-hour post-dose observation period to check for injection site reaction and/or adverse reactions.
  Interventions: Drug: CpG1018
- CpG 1018 0.5 mg/kg (Experimental): 3 injections at Day 1, Week 4, and Week 8.
  Treatment administered as morning injection of dose 0.5 mg/kg, followed by 1-hour post-dose observation period to check for injection site reaction and/or adverse reactions.
  Interventions: Drug: CpG1018
- Placebo (Placebo Comparator): 3 injections of sterile saline at Day 1, Week 4, and Week 8, followed by 1-hour post-dose observation period to check for injection site reaction and/or adverse reactions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CpG1018 — 0.1 mg/kg dose administered via subcutaneous injection.
  TLR9 agonist supplied by Dynavax Technologies Inc.
  Arms: CpG 1018 0.1 mg/kg
Drug: CpG1018 — 0.25 mg/kg dose administered via subcutaneous injection.
  TLR9 agonist supplied by Dynavax Technologies Inc.
  Arms: CpG 1018 0.25 mg/kg
Drug: CpG1018 — 0.5 mg/kg dose administered via subcutaneous injection.
  TLR9 agonist supplied by Dynavax Technologies Inc.
  Arms: CpG 1018 0.5 mg/kg
Drug: Placebo — Sterile saline injection supplied by the NYU Investigational Pharmacy.
  Arms: Placebo

SUMMARY:
This single-center, double-blind, placebo-controlled study will recruit in total 39 participants with either Mild Cognitive Impairment due to Alzheimer's disease (MCI) or Mild Alzheimer's disease dementia (mild AD). There will be 3 Dose levels. An initial cohort of 13 subjects will be randomized to a Dose level 1 (0.1 mg/kg vs. placebo) lasting 8 weeks. An additional 13 subjects will be recruited and randomized into Dose level 2 (0.25 mg/kg vs. placebo) for 8 weeks and 13 subjects for the last Dose level 3 (0.5 mg/kg vs. placebo) for 8 weeks. The primary objective will be to assess safety and tolerability of CpG 1018.

ELIGIBILITY:
Inclusion Criteria:

1. 65-85 years of age
2. MCI due to AD or mild AD dementia per NIA-AA specified criteria published in 2018
3. Montreal Cognitive Assessment (MoCA) score ≥17 AND;
4. Positive Florbetaben PET amyloid scan, or other positive PET amyloid scan performed within one year of study enrollment
5. Must be able to provide consent or assent (If applicable).
6. Must be willing and able to participate in all study related procedures.
7. Must have a reliable study partner to provide information on the subject's cognitive and functional status. Study partner must have sufficient contact with the subject, as determined by the PI, and be available to accompany the subject to clinic visits or by phone.

Exclusion Criteria:

1. History of psychiatric illness (e.g. hallucinations, major depression, suicidal ideation or delusions) that could interfere with completion of study related procedures as determined by PI
2. History of autoimmune disorders or antibody-mediated disease, severe asthma, or other serious infection or systemic illness, as determined by PI
3. Use of corticosteroids or immunosuppressive drugs within 30 days of study entry
4. History of splenectomy
5. Renal impairment
6. Use of chloroquine within 8 weeks of study entry
7. Inability to undergo MRI imaging
8. History of TIA, stroke or seizures within 12 months of screening
9. Any neurological condition other than AD that could contribute to cognitive impairment (including related to possible "long COVID") as determined by PI
10. Participation in any other current AD investigational interventional trial
11. Current use of an anti-coagulant
12. Current use of drugs that are major substrates of cytochrome P450 (CYP) enzyme 1A2
13. Recent exposure to COVID-19 infection within 14 days or recent onset of symptoms within 14 days that may be related to COVID-19 infection

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of Patient-Reported Adverse Events (AEs) | Up to Week 18
  AEs defined as any symptom, sign, illness or experience that develops or worsens in severity during the course of the study.
Percentage of Participants with Rheumatoid Factor (RF) Confirmed by Autoimmunity Marker Screening Test Result | Up to Week 18
  Evaluation of RF in patient blood samples at Baseline, Day 56, Week 14 and Week 18.
Percentage of Participants with Antinuclear Antibody (ANA) Confirmed by Autoimmunity Marker Screening Test Result | Up to Week 18
  Evaluation of ANA in patient blood samples at Baseline, Day 56, Week 14 and Week 18.
Percentage of Participants with Antineutrophil Cytoplasmic Antibody (ANCA) Confirmed by Autoimmunity Marker Screening Test Result | Up to Week 18
  Evaluation of ANCA in patient blood samples at Baseline, Day 56, Week 14 and Week 18.
Percentage of Participants with Amyloid-Related Imaging Abnormalities-Haemosiderin (ARIA-H) Confirmed by Magnetic Resonance Imaging (MRI) | Up to Week 14
  Evaluation of ARIA-H at Baseline and Week 14 using 3T PET/MR Siemens Biograph system.
Percentage of Participants with Amyloid-Related Imaging Abnormalities-Edema (ARIA-E) Confirmed by Magnetic Resonance Imaging (MRI) | Up to Week 14
  Evaluation of ARIA-E at Baseline and Week 14 using 3T PET/MR Siemens Biograph system.

SECONDARY OUTCOMES:
Change in AD Assessment Scale Cognitive Subscale (ADAS-Cog-13) Scores | Baseline, Week 18
  13-item self-assessment measuring levels of cognitive and non-cognitive dysfunctions from mild to severe. Total scores range from 0 to 85. Lower scores indicate greater cognitive performance. A decrease in scores indicates cognitive performance improved during the observational period.
Change in AD Cooperative Study-Activities of Daily Living Inventory, Mild Cognitive Impairment version (ADCS-ADL-MCI) Scores | Baseline, Week 18
  18-item questionnaire measuring a participant's basic and instrumental activities of daily living over the previous month. Total scores range from 0-53, where higher scores indicate greater competence in performing activities. An increase in scores indicates competence increased during the observational period.
Change in Columbia-Suicide Severity Rating Scale (C-SSRS) Scores | Baseline, Week 18
  C-SSRS systematically tracks suicidal ideation and behavior. The total score range is 0 (no ideation is present) to 5 (active suicidal ideation with specific plan and intent). A decrease in scores indicates suicidal ideation and behavior decreased during the observational period.
Change in Global Clinical Dementia Rating (CDR-Global) | Baseline, Week 18
  5-point questionnaire assessing six domains of cognitive and functional performance applicable to Alzheimer's disease and related dementias: Memory, Orientation; Judgement & Problem Solving; Community Affairs; Home & Hobbies; and Personal Care. Higher scores indicate greater severity of dementia: 0= Normal, 0.5=very mild dementia, 1=mild dementia, 2=moderate dementia, 3=severe dementia.
Change in Montreal Cognitive Assessment (MoCa) Score | Baseline, Week 18
  30-item assessment of global cognitive function. Total scores range from 0 to 30, with higher scores indicating greater cognitive function. Scores of 26 and higher are consider to be normal. An increase in scores indicates cognitive function increased during the observational period.
Change in Plasma Amyloid Biomarker Concentration | Baseline, Week 18
  Amyloid biomarker concentration detected via plasma analysis.
Change in Cerebral Spinal Fluid (CSF) Amyloid Biomarker Concentration | Baseline, Week 18
  Amyloid biomarker concentration detected via CSF analysis.
Change in Plasma Tau Biomarker Concentration | Baseline, Week 18
  Tau biomarker concentration detected via plasma analysis.
Change in CSF Tau Biomarker Concentration | Baseline, Week 18
  Tau biomarker concentration detected via CSF analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Arjun Masurkar, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Alok.Vedvyas@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Alok.Vedvyas@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.